CLINICAL TRIAL: NCT01425372
Title: A Prospective Study to Evaluate the Immune Response of UK Infants Receiving the 13-valent Pneumococcal Conjugate Vaccine as Part of Their Routine Primary Immunisation Schedule at 2 and 4 Months
Brief Title: Evaluating Vaccine Responses in Healthy Infants Receiving Their Routine Primary Immunisation According to the Accelerated United Kingdom Schedule at 2, 3 and 4 Months
Acronym: P13UK
Status: Completed | Type: Observational
Sponsor: Prof. Elizabeth Miller (Other Government)
Responsible Party: Sponsor-Investigator, Prof. Elizabeth Miller, Consultant Epidemiologist, Public Health England
Organization: Public Health England (Other Government)
Other Study IDs: P13UK
Record Dates: First submitted 2011-08-26; First posted 2011-08-30 (Estimated); Last update posted 2019-03-22 (Actual); Status verified 2018-08

CONDITIONS: Streptococcus Pneumoniae
Keywords: vaccine; pneumococcal conjugate vaccine; immune responses; primary immunisation; Vaccine responses to primary immunisation in the UK

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Streptococcus pneumoniae is a major cause of serious bacterial infections, particularly among young children. Over 30 different types of the pneumococcus germ can cause invasive disease, but 7 types (namely serotypes 4, 6B, 9V, 14, 18C, 19F and 23F) are responsible for around 75% of cases in young children. A pneumococcal conjugate vaccine against these 7 serotypes (PCV7; Prevenar ®, Wyeth Vaccines) was introduced into the UK national immunisation programme in September 2006 and has resulted in a rapid reduction in pneumococcal disease caused by the 7 serotypes among both vaccinated children and older unvaccinated children and adults through herd immunity. By 2009, over half of all invasive pneumococcal cases in young children were caused by six other pneumococcal serotypes (1, 3, 5, 6A, 7F and 19A) that are included in a newly licensed 13 valent pneumococcal vaccine (PCV13; Prevenar 13®, Wyeth Vaccines). In April 2010, PCV13 replaced PCV7 in the UK immunisation programme with the aim of further reducing cases of invasive pneumococcal disease. The antibody responses induced by the 7 serotypes in both PCV13 and PCV7 have been shown to be comparable, but the protection offered by the additional 6 serotypes in PCV13 merits further study. Also, it is possible that the use of PCV13 instead of PCV7 may interfere with immune responses to other vaccines, such as Haemophilus influenzae serotype b (Hib), which are given to infants at the same time as PCV13. The proposed study will aim to collect one blood sample from infants after they receive their routine vaccinations at 2, 3 and 4 months in order to their measure immune responses to routine vaccines. The investigators hope that their results will help us better understand the added protection offered by the 13valent pneumococcal vaccine and ensure that children are adequately protected by the other vaccines they receive.

DETAILED DESCRIPTION:
This study will aim to prospectively recruit infants in the first 6 months of life who are either due to receive or in the process of receiving their routine infant immunisation and request one blood sample one month after completing their primary immunisation schedule, which will be at around 5 months of age, if they fulfil the inclusion criteria for the study.

NUMBER OF SUBJECTS AND DURATION OF STUDY

A total of 200 infants will be recruited in two centres - Hertfordshire and Gloucestershire.

ELIGIBILITY:
Inclusion Criteria:

Male or female infants born at term (at least 37 weeks gestation) aged <6 months:

1. With written informed consent obtained from the parent or legal guardian of the infant to participate in the study and to allow the infant's General Practitioner (GP) to be informed of participation in the study and be contacted, if required, for confirmation of the vaccination history
2. Who have received all their primary immunisations in the 1st 6 months of life, including:

   * 3 doses of Pediacel®
   * 2 doses of Prevenar13®, with the 1st dose given at 6-12 weeks of age and the 2nd dose at 8-12 weeks after the 1st dose
   * 2 doses of any MenC vaccine
3. Do not fulfil any of the Exclusion Criteria

Exclusion Criteria:

Participant may not be included in the study if any of the following apply:

1. History of invasive Haemophilus influenzae serotype b (Hib), pneumococcal or meningococcal disease
2. Confirmed or suspected immunosuppressive or immunodeficient condition (including HIV)
3. Bleeding disorders and/or prolonged bleeding time
4. Major congenital defects or chronic disease
5. Premature birth (<37 weeks gestation at birth)

Max Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy infants who have received their primary immunisation schedule at appropriate intervals
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2010-11; Primary Completion 2012-05 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
1. To determine the proportion of infants with pneumococcal serotype-specific IgG antibody concentrations ≥0.35 μg/ml for the 13 serotypes included in Prevenar13 at one month after completion of primary immunisation | 24 months

SECONDARY OUTCOMES:
1. To determine the geometric mean concentrations (GMCs) of pneumococcal serotype-specific IgG antibody concentrations for each of the 13 serotypes in Prevenar13 one month after primary immunisation | 24 months
2. To determine, using a functional opsonophagocytic assay (OPA), the proportion of infants with geometric mean titres (GMT) ≥1:8 for the 13 serotypes in Prevenar13 one month after primary immunisation | 24 months
3. To determine serum bactericidal assay (SBA) titres with 95%CI for MenC and the proportion of infants achieving SBA titres ≥8 or ≥128 one month after primary immunisation | 24 months
4. To determine Hib GMC with 95%CI and proportions of infants with Hib antibody concentrations ≥0.15 μg/ml or ≥1.0 μg/ml one month after primary immunisation | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Coates, PhD, Study Chair — Public Health England
Locations (1):
- Multiple GP surgeries, Hertfordshire and Gloucstershire, United Kingdom

REFERENCES:
- [Background] Andrews NJ, Waight PA, Burbidge P, Pearce E, Roalfe L, Zancolli M, Slack M, Ladhani SN, Miller E, Goldblatt D. Serotype-specific effectiveness and correlates of protection for the 13-valent pneumococcal conjugate vaccine: a postlicensure indirect cohort study. Lancet Infect Dis. 2014 Sep;14(9):839-46. doi: 10.1016/S1473-3099(14)70822-9. Epub 2014 Jul 17. PMID 25042756
- [Result] Ladhani SN, Andrews NJ, Waight P, Hallis B, Matheson M, England A, Findlow H, Bai X, Borrow R, Burbidge P, Pearce E, Goldblatt D, Miller E. Interchangeability of meningococcal group C conjugate vaccines with different carrier proteins in the United Kingdom infant immunisation schedule. Vaccine. 2015 Jan 29;33(5):648-55. doi: 10.1016/j.vaccine.2014.12.018. Epub 2014 Dec 12. PMID 25510388
- See also: Published study results — https://www.ncbi.nlm.nih.gov/pubmed/25510388?dopt=Abstract
- See also: Published study results — https://www.ncbi.nlm.nih.gov/pubmed/25042756